CLINICAL TRIAL: NCT04364373
Title: D2 vs D3 Lymph Node Dissection for Left Colon Cancer: Multicenter Randomize Control Trial (DILEMMA)
Brief Title: D2 vs D3 Lymph Node Dissection for Left Colon Cancer
Acronym: DILEMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Society of Colorectal Surgeons (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other); G.V. Bondar Republican Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2020-04-01; First posted 2020-04-28 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colon Cancer
Keywords: D2; D3; lymph node dissection; complete mesocolic excision; left colon cancer; CME
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 lymph node dissection (Active Comparator): For tumours in splenic flexure and proximal and mid part of descending colon lymph nodes 232 and 231 will be removed.
  For tumours in distal part of descending colon and proximal sigmoid lymph nodes 231, 232 and partially 241, 242 (considering variation of the feeding artery) will be removed.
  For tumours in the mid part of sigmoid colon lymph nodes 241, 242 will be removed.
  For tumours in the rectosigmoid junction 251, 252 groups of the lymph node will be removed.
  Interventions: Procedure: Left colon resection; Procedure: Sigmoid colon resection; Procedure: Distal sigmoid colon resection or anterior resection
- D3 lymph node dissection (Experimental): For tumours in splenic flexure and proximal and mid part of descending colon lymph nodes 232, 231 and 253 will be removed.
  For tumours in distal part of descending colon and proximal sigmoid lymph nodes 231, 232 and 253 and partially 241, 242 (considering variation of the feeding artery) will be removed.
  For tumours in the mid part of sigmoid colon lymph nodes 241, 242 and 253 will be removed.
  For tumours in the rectosigmoid junction 251, 252 and 253 groups of the lymph node will be removed.
  Interventions: Procedure: Left colon resection; Procedure: Sigmoid colon resection; Procedure: Distal sigmoid colon resection or anterior resection

INTERVENTIONS:
Procedure: Left colon resection — This procedure is performed for tumours in splenic flexure and proximal and descending colon.
  Left colic artery is divided at its origin. Sigmoid arteries and superior rectal arteries are preserved. Inferior mesenteric vein is divided at the lower border of the pancreas. The colon is divided about 10 cm proximal and distal to the tumour. Mesocolic fascia is preserved and the length of the "vessel trunk" of the mesocolon corresponds to the level of lymph node dissection. After removal of the resected colonic segment a handsewn or stapler end-to-end or side-to-side colonic anastomosis is performed.
Procedure: Sigmoid colon resection — This procedure is performed for tumours in sigmoid colon. Corresponding sigmoid arteries are divided at their origin. Left colic artery and superior rectal artery are preserved. Inferior mesenteric vein is divide close to the left colic artery. Proximal and distal margin compose 10 cm from the tumour. Mesocolic fascia is preserved and the length of the "vessel trunk" of the mesocolon corresponds to the level of lymph nodes dissection. After removal of the resected colonic segment a handsewn end-to-end or side-to-side or stapler colonic anastomosis is performed.
Procedure: Distal sigmoid colon resection or anterior resection — This procedure is performed for tumours in distal sigmoid colon or rectosigmoid junction. Superior rectal artery is divided below the origin of left colic artery. Left colic artery is preserved. Inferior mesenteric vein is divide close to the left colic artery. The colon is divided about 10 cm proximal and 5 cm distal to the tumour. Mesocolic fascia is preserved and the length of the "vessel trunk" of the mesocolon corresponds to the level of lymph node dissection. After removal of the resected colonic segment handsewn or stapler colo-rectal anastomosis is performed.

SUMMARY:
The efficiency of the D3 lymph node dissection is still controversial for left colon cancer patients. This study will try find difference in 5-year overall survival between D2 and D3 lymph node dissection. Investigation of the functional and short-term outcomes will clarify safety of the D3 lymph node dissection.

DETAILED DESCRIPTION:
Discussion about optimal type of lymph node dissection in colorectal cancer continues during last 15 years, when in Europe was presented concept of complete mesocolic excision. However, this concepts is very close to Japanese D3 lymph node dissection and in the first view it seems the same but principal differences were found. Japanese concept is partial resection of the bowel according feeding artery (short bowel specimen, long lymphovascular pedicle), opposite European concept is wide resection of the bowel like hemicolectomy or extended hemicolectomy, sigmoidectomy. In complete mesocolic excision anatomical landmarks are still unclear but in Japanese guidelines it has anatomical margins which can standardize this procedure. Also nerve sparing technique around root of inferior mesenteric artery was described. One more difference is in histological examination of the specimen. European concept is to pay more attention to the quality of complete mesocolic excision and less - to the number of investigated lymph nodes. In Japan lymph node extraction is performed by surgical team from the fresh specimen and send to pathologist separately (each group of lymph nodes). Considering the absence of randomized control trials for patients with left colon cancer DILEMMA trial was started using Japanese approach

ELIGIBILITY:
Inclusion Criteria:

1. Agreement of the patient to participate in trial
2. Colon cancer (only adenocarcinoma )
3. The tumor located between the splenic flexure and rectosigmoid junction
4. cT3-Т4а,b
5. cN0-2
6. cM0
7. Tolerance of chemotherapy
8. ASA 1-3

Exclusion Criteria:

1. сТis - Т2, сТ4b (tail of the pancreas, stomach, small bowel, ureter, urinary bladder)
2. Preoperative complications of the tumor (perforation and full bowel 3. obstruction)
3. Previous radiotherapy or chemotherapy
4. Synchronous or metachronous tumors
5. Women during Pregnancy or breast feeding period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1381 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | Up to 5 years post-operatively
  Probability to be alive measured in %, where 100% means that patients have a 100% probability to be alive and 0% means that patients have 0% probability to be alive

SECONDARY OUTCOMES:
5-year disease free survival | Up to 5 years post-operatively
  Probability to be alive with no signs of local or distant recurrence measured in %, where 100% means that patients have a 100% probability to be alive with no signs of local or distant recurrence and 0% means that patients have 0% probability to be alive with no signs of local or distant recurrence
Postoperative sexual dysfunction | Up to 1 year post-operatively
  The rate of ejaculation problems in sexually active men and the rate of decreased vaginal lubricant production in sexually active women, measured in % from the total number of male/female patients
Apical lymph node involvement rate | 1 month after surgery
  The rate of lymph nodes 253 with metastatic cells among all lymph nodes 253, measured in %
Intraoperative complications rate | Day 0
  The rate of any complications within the course of surgery
Early postoperative complications rate | 1-30 days after surgery
  The rate of surgical and infectious complications
Mortality | 0-30 days after surgery
  The rate of death from all causes
Late postoperative complications rate | 30-180 days after surgery
  The rate of surgical and infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tsarkov, Ph.D, Study Director — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Clinic of coloproctology and minimally invasive surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No